CLINICAL TRIAL: NCT02778958
Title: Comparisons of iv Ibuprofen and iv Paracetamol for Postoperative Pain Levels and Opioid Consumption During Bariatric Surgery
Brief Title: Comparisons of iv Ibuprofen and iv Paracetamol During Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, Director of the study, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inonu Medicine Faculty
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
Keywords: bariatric surgery; morbid obesity; nonopioid analgesics
MeSH Terms: conditions — Obesity, Morbid | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibuprofen and morphine (Experimental): iv ibuprofen 800 mg infusion at 30 min before skin incision closed and per 6 hours during postoperative period; iv morphine with patient controlled analgesia (1 mg demand bolus dose, 20 min lockout time)
  Interventions: Drug: ibuprofen
- paracetamol and morphine (Active Comparator): iv paracetamol 1 gram infusion at 30 min before skin incision closed and per 6 hours during postoperative period; iv morphine with patient controlled analgesia (1 mg demand bolus dose, 20 min lockout time)
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — iv paracetamol flakon, 1 gram infusion at 30 min;
  iv morphine with patient controlled analgesia (1 mg demand bolus dose, 20 min lockout time)
  Other Names: Acetaminophen
  Arms: paracetamol and morphine
Drug: ibuprofen — iv ibuprofen flakon, 800 mg;
  iv morphine with patient controlled analgesia (1 mg demand bolus dose, 20 min lockout time)
  Other Names: İntrafen
  Arms: ibuprofen and morphine

SUMMARY:
The aim of this study is to evaluate and to compare the effectiveness of iv ibuprofen and iv paracetamol during bariatric surgery.

DETAILED DESCRIPTION:
Evaluation of effectiveness of iv ibuprofen and iv paracetamol on postoperative pain, opioid consumption, and side effects in morbidly obese patients undergoing bariatric laparoscopic surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic sleeve gastrectomy and gastric by-pass surgery

Exclusion Criteria:

* Hepatic disfunction,
* Renal failure (creatinine > 3 mg/dL,creatinin clearance < 60 mL/dk or urine out-put < 500 mL/day ) or a history of dialysis 28 days before surgery,
* A history of gastrointestinal bleeding or bleeding diathesis 6 weeks before surgery, therapeutic dose of anticoagulation therapy (except subcutaneous heparin prophylactic dose),
* Angiotensin converting enzymes inhibitor or antihypertensive combination with furosemide,
* A history of opioid addiction or opioid tolerance
* Allergy to study drugs,
* Noncooperative patients for pain assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Opioid (morphine) consumption | First 24 hours during postoperative period
  iv morphine patient controlled analgesia for multimodal analgesia

SECONDARY OUTCOMES:
Postoperative pain level | First 24 hours during postoperative period
  Visual analog scale for evaluation of postoperative pain levels

OTHER OUTCOMES:
Side effects | First 24 hours during postoperative period
  Side effects of study drugs and opioids

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Erdogan Kayhan, MD, Principal Investigator — Associated Professor Doctor Gulay ERDOGAN KAYHAN
Locations (1):
- Inonu University Faculty of Medicine Department of Anesthesiology and Reanimation, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488